CLINICAL TRIAL: NCT01124409
Title: Randomised Clinical Phase III Study of Radiotherapy Dose, Volume Evaluation for 3DCRT Versus IGRT and Analysis of Early Response in Head and Neck Squamous Cell Carcinoma
Brief Title: Evaluation of 3DCRT Versus IGRT and Analysis of Early Response in Head and Neck Cancer.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: DR.SUJITH KUMAR MULLAPALLY, ALL INDIA INSTITUTE OF MEDICAL SCIENCES
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3DIGHNC
Record Dates: First submitted 2010-05-13; First posted 2010-05-17 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: HEAD AND NECK CANCER; CARCINOMA OROPHARYNX; CARCINOMA PYRIFORM SINUS; CARCINOMA LARYNX
Keywords: IGRT; 3DCRT; EPID; CBCT; HNSCC
MeSH Terms: conditions — Head and Neck Neoplasms; Laryngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3DCRT with EPID (Active Comparator): this patients randomised to this arm will be planned by 3DCRT and during treatment setup error will be identified and corrected by weekly EPID if error >3mm.Weekly CBCT will be done for this arm to note the setup error but will not be corrected.
  Interventions: Radiation: EPID Verification
- IGRT with CBCT (Active Comparator): The patients randomised to this arm will be planned by 3DCRT and set up error during RT will be verified by CBCT and error corrected if >3mm.Weekly EPID will be done for setup error documentation but no correction based on EPID in this arm.
  Interventions: Radiation: CBCT verification

INTERVENTIONS:
Radiation: EPID Verification — Set up error verification and correction by EPID
  Other Names: EPID; 3DCRT; HNSCC
  Arms: 3DCRT with EPID
Radiation: CBCT verification — Setup error verification and correction by CBCT
  Other Names: CBCT; IGRT; HNSCC
  Arms: IGRT with CBCT

SUMMARY:
This study aims to study the impact image guided radiotherapy with Cone beam CT will have on the outcomes(toxicities and response) of head and neck cancer when compared to 3D conformal radiotherapy without CBCT based setup error verification.Also,the various dosimetric variations in Adaptive RT will be studied.

DETAILED DESCRIPTION:
Aims and Objectives

1. To assess the patient's radiation dose planning for GTV, CTV and PTV for primary and nodal regions and derive comparison between IGRT and 3D-CRT.
2. To assess the dosimetric variation in different phases of adaptive RT due to changes in tumor shape and volume during the course of entire treatment in IGRT arm in head and neck cancer patients.
3. To evaluate the optimal setup correction methodology using planar (EPID) and volumetric images (CBCT) in HNSCC between 3D-CRT and IGRT treatment delivery respectively.
4. To compare the early tumour response and acute and chronic radiation morbidities between IGRT and 3D-CRT.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically proven cases of Carcinoma Oropharynx,Larynx,Hypopharynx, stages T1-4 N0-2a M0
* Informed Consent
* KPS score > 70

Exclusion Criteria:

* Uncontrolled medical comorbidity
* Not ready for follow up
* Previous cancer directed therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-12; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
compare the early tumour response between 3DCRT and IGRT in head and neck cancer. | Assessment at post RT week, 1 month after completion of RT and 6 month after completion of RT. Final assessment of last recruited patient is anticipated to be by AUGUST 2011
  The advent of CBCT has increased the verification of Radiation treatment delivery but whether it leads to significant change in tumour response or toxicities when compared to 3D Conformal Radiotherapy without CBCT verification is not known.This study will give insights into this question.

SECONDARY OUTCOMES:
To assess and compare early and late toxicities between 3DCRT and IGRT in head and neck cancer | assessment of acute and chronic toxicities of the last recruited patient anticipated to be by March 2011
  Assessment will be done by RTOG scoring criteria
To find out the different doses received by target and organs at risk during the various phases of adaptive RT. | last measurement by AUG 2011

CONTACTS AND LOCATIONS:
Overall Officials: BIDHU K MOHANTI, MD, Study Chair — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, New Delhi, India